CLINICAL TRIAL: NCT00550771
Title: Randomized Phase II Multinational Trial to Evaluate the Safety of Two Chemotherapy Plus Trastuzumab Regimens as Adjuvant Therapy in Patients With HER2-positive Breast Cancer: Caelyx + Cyclophosphamide + Trastuzumab (C+C+H) or Doxorubicin + Cyclophosphamide (A+C), Each Followed by Paclitaxel + Trastuzumab (T+H) BACH
Brief Title: Phase II Trial to Compare the Safety of Two Chemotherapy Plus Trastuzumab Regimens as Adjuvant Therapy for HER2-positive Breast Cancer (Study P05048)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05048
Record Dates: First submitted 2007-10-29; First posted 2007-10-30 (Estimated); Results first posted 2011-10-03 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-05

CONDITIONS: Breast Neoplasm
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Cyclophosphamide; Paclitaxel; Trastuzumab; 1-dodecylpyridoxal; liposomal doxorubicin

ARMS (2):
- Doxorubicin Based Regimen (Active Comparator)
  Interventions: Drug: doxorubicin, cyclophosphamide, paclitaxel, trastuzumab
- Pegylated Liposomal Doxorubicin (PLD) Based Regimen (Experimental)
  Interventions: Drug: PLD, cyclophosphamide, trastuzumab, paclitaxel

INTERVENTIONS:
Drug: doxorubicin, cyclophosphamide, paclitaxel, trastuzumab — doxorubicin 60 mg/m^2 IV push + cyclophosphamide 600 mg/m^2 IV over 30-90 minutes given every 21 days for 4 courses (12 weeks) followed by Paclitaxel 80 mg/m^2 IV over 60 minutes with trastuzumab 2 mg/kg IV over 30 minutes (first administration 4 mg/kg IV over 90 minutes) given weekly for 12 weeks (4 courses)
  Arms: Doxorubicin Based Regimen
Drug: PLD, cyclophosphamide, trastuzumab, paclitaxel — PLD 35 mg/m^2 IV over 60 minutes + cyclophosphamide 600 mg/m^2 IV over 30-90 minutes given every 21 days + trastuzumab 2 mg/kg IV over 30 minutes (first dose 4 mg/kg IV over 90 minutes) given once weekly for 4 courses (12 weeks) followed by Paclitaxel 80 mg/m^2 IV over 60 minutes with trastuzumab 2 mg/kg IV over 30 minutes given weekly for 12 weeks (4 courses)
  Other Names: pegylated liposomal doxorubicin (SCH 200746)
  Arms: Pegylated Liposomal Doxorubicin (PLD) Based Regimen

SUMMARY:
The purpose of this study is to compare the incidence of cardiac dysfunction in subjects with human epidermal growth factor receptor 2 (HER2) positive breast cancer treated with either doxorubicin or pegylated liposomal doxorubicin (PLD), both in combination with trastuzumab.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with operable, node-positive or high-risk node-negative (see #3 below) HER2-positive breast carcinoma are eligible for the study, provided they satisfy the following criteria.

  * Subjects must demonstrate willingness to and be able to participate in the study and to adhere to dose and visit schedules
  * Subjects must be of female gender and >= 18 years of age
  * Subjects must have been diagnosed with operable, histologically confirmed adenocarcinoma of the breast with no clinical or radiological evidence of metastatic disease but with otherwise high or intermediate risk tumor characteristics:

    * node-positive: T1-3, N1-2, M0 (level of T [tumor involvement], N [lymph node involvement], & M [matastases]) OR
    * node-negative AND at least one of the following features:

      * Tumor >2 cm or
      * Tumor >1 cm and

        * Negative estrogen receptor/progesterone receptor (ER/PR) or
        * Malignancy Grade 2-3 or
        * Presence of peritumoral vascular invasion or
        * Age <35 years
  * HER2-positive by fluorescence in situ hybridization (FISH)(with gene amplification) or 3+ using

immunohistochemistry

* Subjects must have had complete resection (R0) of the primary tumor and axillary lymph nodes (or must have negative sentinel node[s])
* Baseline left ventricular ejection fraction (LVEF) by multiple gated acquisition (MUGA) scan or echocardiogram (ECHO) >=55%
* Easter Cooperative Oncology Group (ECOG)-performance status of 0-1
* Adequate postoperative bone marrow function with neutrophils >=1.5 x 10^9/l, platelets >=100 x 10^9/l and hemoglobin >= lower limit of normal (LLN)
* Adequate renal function: calculated creatinine clearance >=50 ml/min
* Adequate postoperative liver function with a total bilirubin < upper limit of normal (ULN), alkaline phosphatase <2.5 times the ULN and aspartate aminotransferase (AST) <1.5 times the ULN
* Subjects must be free of any clinically relevant disease that would, in the principal investigator's and/or sponsor's opinion, interfere with the conduct of the study or study evaluations
* Subjects of childbearing potential (including women who are less than one year postmenopausal and will be sexually active during the study) must agree to use a medically accepted method of contraception, while receiving protocol-specified medication and for 30 days (or as per local requirements) after stopping the medication or be surgically sterilized prior to screening
* Subjects must be able to provide written informed consent

Exclusion Criteria:

* Subject who meets any of the following exclusion criteria will be disqualified from participation in the study:

  * Clinical or radiological evidence of metastatic disease
  * Prior radiotherapy, chemotherapy or biotherapy for the currently diagnosed breast cancer prior to randomization
  * Clinically significant pericardial effusion
  * Serious cardiac illness including, but not confined to

    * history of documented congestive heart failure
    * history of any form of cardiomyopathy or active treatment for any form of cardiomyopathy
    * history of angina pectoris or documented transmural myocardial infarction, or active angina pectoris requiring medication
    * serious ventricular arrhythmias requiring medication or implantable cardioverter-defibrillator (ICD) therapy, uncontrolled supraventricular arrhythmias
    * clinically significant valvular disease
    * poorly controlled arterial hypertension (systolic blood pressure (BP) >180 mmHg, diastolic BP >100 mmHg)
  * Sensory/motor neuropathy > grade 2 as defined by National Cancer Institure - Common Toxicity Criteria (NCI-CTC)
  * Pregnancy, or intending to become pregnant during the study
  * Nursing (breastfeeding) or intending to be nursing during the study
  * Any of the following clinical conditions:

    * Chronic obstructive pulmonary disease, requiring chronic treatment
    * Clinically significant active infections
    * A history of a psychological illness of condition, preventing the subject to understand the requirements of the study
    * Unstable regulation of diabetes mellitus
  * A situation or condition that, in the opinion of the investigator, may interfere with optimal participation in the study
  * Is on staff, affiliated with, or a family member of the staff personnel directly involved with this study
  * Usage of any investigational product within 30 days prior to enrollment
  * Participation in any other interventional clinical study involving drug, device or biological. This would not prohibit the patient from participating in a quality of life (QOL), questionnaire, blood collection, or observational study.
  * Allergy to or sensitivity to the study drug or its excipients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2007-07-16 (Actual); Primary Completion 2010-08-23 (Actual); Study Completion 2010-08-23 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Rayson D, Suter TM, Jackisch C, van der Vegt S, Bermejo B, van den Bosch J, Vivanco GL, van Gent AM, Wildiers H, Torres A, Provencher L, Temizkan M, Chirgwin J, Canon JL, Ferrandina G, Srinivasan S, Zhang L, Richel DJ. Cardiac safety of adjuvant pegylated liposomal doxorubicin with concurrent trastuzumab: a randomized phase II trial. Ann Oncol. 2012 Jul;23(7):1780-8. doi: 10.1093/annonc/mdr519. Epub 2011 Nov 4. PMID 22056854

RESULTS

PARTICIPANT FLOW:
Groups:
- Pegylated Liposomal Doxorubicin (PLD) Based Regimen: PLD 35 mg/m^2 IV over 60 minutes + cyclophosphamide 600 mg/m^2 IV over 30-90 minutes given every 21 days + trastuzumab 2 mg/kg IV over 30 minutes (first dose 4 mg/kg IV over 90 minutes) given once weekly for 4 courses (12 weeks) followed by Paclitaxel 80 mg/m^2 IV over 60 minutes with trastuzumab 2 mg/kg IV over 30 minutes given weekly for 12 weeks (4 courses)
- Doxorubicin Based Regimen: doxorubicin 60 mg/m^2 intravenous (IV) push + cyclophosphamide 600 mg/m^2 IV over 30-90 minutes given every 21 days for 4 courses (12 weeks) followed by Paclitaxel 80 mg/m^2 IV over 60 minutes with trastuzumab 2 mg/kg IV over 30 minutes (first administration 4 mg/kg IV over 90 minutes) given weekly for 12 weeks (4 courses)
Period: Overall Study
Arm/Group | Pegylated Liposomal Doxorubicin (PLD) Based Regimen | Doxorubicin Based Regimen
Started | 121 | 60
Completed | 104 | 50
Not Completed | 17 | 10
Not completed — Adverse Event | 11 | 3
Not completed — Discontinued for study-related reasons | 0 | 1
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol Violation | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pegylated Liposomal Doxorubicin (PLD) Based Regimen | Doxorubicin Based Regimen | Total
Number analyzed (Participants) | 120 | 59 | 179
Age, Continuous [Mean (Standard Deviation); unit: years] — Age information was for the intent-to-treat (ITT) population (n=59 for doxorubicin arm, n=120 for PLD arm). ITT was defined as all participants who were randomized and received at least 1 dose of any study medication.
  years | 50.2 (10.97) | 52.5 (9.32) | 50.9 (10.49)
Sex: Female, Male [Count of Participants; unit: Participants] — ITT population.
  Participants
    Female | 120 | 59 | 179
    Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Cardiac Events (Level 1 or 2), or Inability to Administer Trastuzumab Either During the 8 Cycles of Chemotherapy or According to Package Insert for a Total Duration of 1 Year
Description: Cardiac events defined as:
  Level 1: Cardiac death due to heart failure (HF), myocardial infarction or arrhythmia, or probable cardiac death defined as sudden, unexpected death within 24 hours of a definite or probable cardiac event, or severe symptomatic HF, concomitant with a left ventricular ejection fraction (LVEF) drop of >10 percentage points from baseline and to ≤50% LVEF
  Level 2: Asymptomatic systolic dysfunction or mildly symptomatic HF concomitant with an LVEF drop of >10 percentage points from baseline and to <50% LVEF; the LVEF drop was to have been confirmed within 3-4 weeks.
Time Frame: 8 cycles of chemotherapy and subsequently one year of planned trastuzumab treatment
Population: ITT, defined as all participants who were randomized and received at least 1 dose of any study medication.
  Each participant could not contribute more than 1 event.
Measure: Number; unit: Participants
Arm/Group | Pegylated Liposomal Doxorubicin (PLD) Based Regimen | Doxorubicin Based Regimen
Number analyzed (Participants) | 120 | 59
Participants | 5 | 11

2. Secondary Outcome: Number of Participants Who Experienced Cardiac Events (Level 1 or 2) or Inability to Administer Trastuzumab During the 8 Cycles of Chemotherapy
Description: as for outcome 1
Time Frame: During the 8 courses of chemotherapy
Population: ITT, defined as all participants who were randomized and received at least 1 dose of any study medication.
Measure: Number; unit: Participants
Arm/Group | Pegylated Liposomal Doxorubicin (PLD) Based Regimen | Doxorubicin Based Regimen
Number analyzed (Participants) | 120 | 59
Participants
  Level 1 Cardiotoxicity | 1 | 0
  Level 2 Cardiotoxicity | 1 | 3
  Inability to Administer Trastuzumab | 0 | 0

3. Secondary Outcome: Number of Participants Who Experienced Cardiac Events (Level 1 or 2) or Inability to Administer Trastuzumab During 1 Year of Trastuzumab Therapy
Description: as for outcome 1
Time Frame: During 1 year of trastuzumab therapy
Population: ITT, defined as all participants who were randomized and received at least 1 dose of any study medication.
Measure: Number; unit: Participants
Arm/Group | Pegylated Liposomal Doxorubicin (PLD) Based Regimen | Doxorubicin Based Regimen
Number analyzed (Participants) | 116 | 52
Participants
  Level 1 Cardiotoxicity | 1 | 0
  Level 2 Cardiotoxicity | 4 | 10
  Inability to Administer Trastuzumab | 4 | 8

4. Secondary Outcome: Number of Participants Who Survived Without Relapse
Description: Relapse-free survival would have been determined by Kaplan-Meier method.
  This was not calculated, since the 2 year follow-up was curtailed.
Time Frame: Approximately 2 years
Arm/Group | Pegylated Liposomal Doxorubicin (PLD) Based Regimen | Doxorubicin Based Regimen
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | PLD Based Regimen | Doxorubicin Based Regimen
Serious Adverse Events (participants affected / at risk) | 20/120 | 7/59
Other Adverse Events (participants affected / at risk) | 115/120 | 58/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLD Based Regimen (N=120) | Doxorubicin Based Regimen (N=59)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 5 (6) | 4 (5)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
ATRIAL THROMBOSIS (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 1 (1) | 1 (1)
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0)
PLEUROPERICARDITIS (Cardiac disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRIC ULCER PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 2 (2)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 2 (2)
INFLUENZA LIKE ILLNESS (General disorders) | 1 (1) | 0 (0)
MALAISE (General disorders) | 0 (0) | 2 (2)
MUCOSAL INFLAMMATION (General disorders) | 0 (0) | 1 (1)
PAIN (General disorders) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 7 (9) | 2 (2)
CELLULITIS (Infections and infestations) | 1 (1) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 1 (1) | 0 (0)
DEVICE RELATED SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
LOCALISED INFECTION (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
UROSEPSIS (Infections and infestations) | 0 (0) | 1 (1)
LETHARGY (Nervous system disorders) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLD Based Regimen (N=120) | Doxorubicin Based Regimen (N=59)
ANAEMIA (Blood and lymphatic system disorders) | 6 (10) | 6 (8)
LEUKOPENIA (Blood and lymphatic system disorders) | 8 (18) | 4 (16)
LYMPHOPENIA (Blood and lymphatic system disorders) | 2 (12) | 3 (3)
NEUTROPENIA (Blood and lymphatic system disorders) | 27 (72) | 26 (37)
PALPITATIONS (Cardiac disorders) | 12 (17) | 4 (7)
DRY EYE (Eye disorders) | 3 (3) | 4 (4)
LACRIMATION INCREASED (Eye disorders) | 11 (12) | 6 (6)
ABDOMINAL PAIN (Gastrointestinal disorders) | 8 (13) | 7 (10)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 8 (8) | 7 (10)
CONSTIPATION (Gastrointestinal disorders) | 31 (45) | 20 (38)
DIARRHOEA (Gastrointestinal disorders) | 34 (65) | 17 (33)
DRY MOUTH (Gastrointestinal disorders) | 1 (1) | 3 (3)
DYSPEPSIA (Gastrointestinal disorders) | 24 (35) | 4 (5)
HAEMORRHOIDS (Gastrointestinal disorders) | 6 (7) | 4 (5)
NAUSEA (Gastrointestinal disorders) | 63 (100) | 35 (70)
STOMATITIS (Gastrointestinal disorders) | 28 (41) | 13 (18)
VOMITING (Gastrointestinal disorders) | 27 (37) | 13 (22)
ASTHENIA (General disorders) | 30 (72) | 11 (27)
CHEST PAIN (General disorders) | 7 (8) | 2 (5)
FATIGUE (General disorders) | 51 (102) | 36 (71)
INFLUENZA LIKE ILLNESS (General disorders) | 3 (5) | 4 (4)
MALAISE (General disorders) | 0 (0) | 4 (9)
MUCOSAL INFLAMMATION (General disorders) | 41 (82) | 16 (21)
OEDEMA (General disorders) | 6 (7) | 5 (7)
OEDEMA PERIPHERAL (General disorders) | 23 (31) | 11 (13)
PAIN (General disorders) | 3 (5) | 3 (3)
PYREXIA (General disorders) | 19 (28) | 10 (14)
HYPERSENSITIVITY (Immune system disorders) | 9 (16) | 3 (3)
NASOPHARYNGITIS (Infections and infestations) | 9 (9) | 6 (6)
SINUSITIS (Infections and infestations) | 1 (1) | 3 (3)
WEIGHT INCREASED (Investigations) | 23 (26) | 14 (23)
DECREASED APPETITE (Metabolism and nutrition disorders) | 29 (38) | 14 (26)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 6 (8) | 7 (12)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 11 (13) | 1 (1)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 5 (9) | 3 (4)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 7 (7) | 4 (6)
MYALGIA (Musculoskeletal and connective tissue disorders) | 20 (26) | 14 (20)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5)
DISTURBANCE IN ATTENTION (Nervous system disorders) | 1 (1) | 3 (3)
DIZZINESS (Nervous system disorders) | 11 (16) | 11 (14)
DYSGEUSIA (Nervous system disorders) | 16 (27) | 8 (15)
HEADACHE (Nervous system disorders) | 18 (30) | 11 (20)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 11 (13) | 8 (12)
NEUROTOXICITY (Nervous system disorders) | 7 (12) | 4 (5)
PARAESTHESIA (Nervous system disorders) | 10 (12) | 5 (6)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 2 (2) | 5 (8)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 16 (35) | 9 (18)
ANXIETY (Psychiatric disorders) | 10 (11) | 2 (2)
DEPRESSION (Psychiatric disorders) | 4 (5) | 4 (4)
INSOMNIA (Psychiatric disorders) | 15 (18) | 7 (9)
DYSURIA (Renal and urinary disorders) | 4 (4) | 4 (4)
COUGH (Respiratory, thoracic and mediastinal disorders) | 19 (24) | 16 (19)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 27 (34) | 12 (21)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 26 (36) | 12 (16)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 10 (13) | 1 (1)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 5 (5)
ALOPECIA (Skin and subcutaneous tissue disorders) | 59 (75) | 45 (55)
DRY SKIN (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (5)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 18 (29) | 2 (3)
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 5 (6) | 6 (6)
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 79 (183) | 3 (3)
RASH (Skin and subcutaneous tissue disorders) | 35 (68) | 6 (8)
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 7 (8) | 0 (0)
FLUSHING (Vascular disorders) | 7 (8) | 2 (2)
HOT FLUSH (Vascular disorders) | 10 (13) | 5 (6)
HYPERTENSION (Vascular disorders) | 4 (5) | 3 (4)

LIMITATIONS AND CAVEATS:
Any follow-up data from this study should be considered with caution as the planned 2-year follow-up was curtailed because of administrative reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The principal investigators (PIs) agree not to publish/publicly present any interim study results without prior sponsor written consent. The PIs further agree to provide 45 days written notice to the sponsor, prior to submission for publication or presentation, to permit the sponsor to review abstracts/manuscripts, which report any study results. The sponsor has the right to review/comment. If the parties disagree, the PIs agree to meet with the sponsor, prior to submission, to discuss/resolve.